CLINICAL TRIAL: NCT05953779
Title: Randomized Controlled Trial for Personalized Need-focused Single-Session Interventions
Brief Title: Personalized Need-focused Single Session Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bar-Ilan University, Israel (Other)
Collaborators: University of California, Berkeley (Other); United States - Israel Binational Science Foundation (Other)
Responsible Party: Principal Investigator, Prof. Eshkol Rafaeli, Professor, Bar-Ilan University, Israel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ER13323
Record Dates: First submitted 2023-03-18; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Depression and/or Anxiety in the Mild-to-moderate Range

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial with 2 conditions: Experimental condition (personalized-selected intervention) and control condition (randomly-selected or standard intervention focused on emotion-regulation).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants and any care provider and study personnel who interact with them will be blind to condition. The PI will utilize a randomization table to allocate participants to condition, and will inform the front-line study personnel and through them, the care provider, regarding which intervention to use without specifying whether it was personalized or randomly-chosen. The outcomes assessor will be blind even to the type of intervention utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Intervention (Experimental): The intervention approach taken in this RCT is focused on unmet psychological needs (predictability, belonging, competence, self-worth, autonomy, and playfulness). For each need, a specific 90-minute intervention has been developed.
  The primary unmet need for each individual will be determined by a conditional entropy algorithm. Simply, the presence versus absence of subjective distress will be measured eight times per day for 30 days. Concurrently, the presence versus absence of need frustration will also be measured eight times per day for 30 days. Utilizing a k-fold cross-validated estimation, conditional entropy will be used to determine the need that best reduces the uncertainty in subjective distress (that is, best explains its presentation probabilistically).
  At both sites, the experimental condition will consist of an algorithmically-chosen intervention. The choice will be made based on data collected during thirty days of ecological momentary assessment.
  Interventions: Behavioral: Clinician-administered Need-focused Single Session Intervention
- Non-personalized Intervention (Active Comparator): The intervention approach taken in this RCT is focused on unmet psychological needs (predictability, belonging, competence, self-worth, autonomy, and playfulness). For each need, a specific 90-minute intervention has been developed.
  At the BIU site, the active control condition will consist of an intervention chosen randomly (out of the six mentioned above).
  At the UCB site, the active control condition will consist of a standard intervention addressing emotion regulation difficulties.
  Interventions: Behavioral: Clinician-administered Need-focused Single Session Intervention

INTERVENTIONS:
Behavioral: Clinician-administered Need-focused Single Session Intervention — All single-session interventions will be 90-minutes in length. At the conclusion of the intervention session, participants will receive suggestions for daily homework practice to complete and a flash drive with a copy of their session audio to review at their discretion. They will also meet with the therapist for a 10-minute remote check-in two weeks following the single session. All interventions include standard psychoeducational components. Both the standard intervention and the specific ones were designed to be broadly efficacious for depression and anxiety symptomatology. The psychosocial needs which serve as the focus of the interventions are derived from motivation and affect regulation models.

SUMMARY:
This is a two-site randomized controlled trial, with two goals. First, the investigators aim to demonstrate that single-session interventions for mild-to-moderate anxiety and depression can generate statistically significant symptom change as a main effect across control and experimental (i.e. personalized) conditions. Second, the investigators hope to establish the additional incremental efficacy of personalization via person-specific intensive longitudinal data collection and analysis.

DETAILED DESCRIPTION:
This is a two-site randomized controlled trial, with two goals. First, the investigators aim to demonstrate that single-session interventions for mild-to-moderate anxiety and depression can generate statistically significant symptom change as a main effect across control and experimental (i.e. personalized) conditions. Second, the investigators hope to establish the additional incremental efficacy of personalization via person-specific intensive longitudinal data collection and analysis.

All single-session interventions will be 90-minutes in length. At the conclusion of the intervention session, participants will receive suggestions for daily homework practice to complete and a flash drive with a copy of their session audio to review at their discretion. Participants will also meet with the therapist for a 10-minute remote check-in two weeks following the single session.

All interventions include standard psychoeducational components. Participants randomized to the personalization arm of the study will be given an intervention matched to their most pressing psychosocial need. Participants randomized to the control condition will receive a standard intervention (at the UCB site) or a randomly selected one (at the BIU site). Both the standard intervention and the specific ones were designed to be broadly efficacious for depression and anxiety symptomatology.

The psychosocial needs which serve as the focus of the interventions are derived from motivation and affect regulation models and include emotional stability, predictability, acceptance, competence, self-esteem, autonomy, and pleasure. The primary unmet need for each individual will be determined by a conditional entropy algorithm. Simply, the presence versus absence of subjective distress will be measured eight times per day for 30 days. Concurrently, the presence versus absence of need frustration will also be measured eight times per day for 30 days. Utilizing a k-fold cross-validated estimation, conditional entropy will be used to determine the need that best reduces the uncertainty in subjective distress (that is, best explains its presentation probabilistically).

ELIGIBILITY:
Inclusion Criterion.

* a score of 5 or above on the Hamilton Rating Scale for Depression (HRSD).

Exclusion Criteria based on Diagnostic Interview for DSM-5 Anxiety, Mood, and Obsessive-Compulsive and Related Disorders (DIAMOND).

* Psychotic Disorders (hallucinations or delusions)
* Past or current mania, current hypo-mania.
* Anorexia Disorder
* Current Obsessive-Compulsive and related Disorders rated as moderate and above.
* Alcohol or drug abuse rated as moderate and above.
* Panic Disorder rated as moderate and above.
* Agoraphobia rated as moderate and above.
* Premenstrual dysphoric disorder rated as moderate and above.
* Current Post-Traumatic Stress Disorder rated as moderate and above.
* binge eating rated as moderate and above.
* Phobia rated as severe and above.
* Somatic symptom disorder rated as severe and above.
* Illness Anxiety Disorder rated as severe and above.
* MDD rated as severe and above.
* GAD rated as severe and above.
* Social Anxiety rated as severe and above.
* Separation anxiety rated as severe and above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-08 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Hamilton-Depression Rating Scale | Change between pre-intervention and 1 month post-intervention
  (Range 0-52, higher scores denote greater depression)
Montgomery-Asberg Depression Rating Scale | Change between pre-intervention and 1 month post-intervention
  (Range 0-60, higher scores denote greater depression)
Hamilton-Anxiety Rating Scale | Change between pre-intervention and 1 month post-intervention
  (Range 0-56, higher scores denote greater anxiety); will be used in lieu of Hamilton-Depression ratings for individuals whose Hamilton-Anxiety scores are higher than their Hamilton-Depression scores.

SECONDARY OUTCOMES:
PHQ-8 | Immediately prior to intervention, and again at 1 and 3 months post-intervention
  (Range 0-24, higher scores denote greater depression)
GAD-7 | Immediately prior to intervention, and again at 1 and 3 months post-intervention
  (Range 0-21, higher scores denote greater anxiety)
DASS | Immediately prior to intervention, and again at 1 and 3 months post-intervention
  (Range 0-63, higher scores denote greater depression, anxiety, and stress)

OTHER OUTCOMES:
PANAS | Up to six weeks prior to intervention, and again at 1 and 3 months post-intervention
  Positive and negative affect schedule (20 items)
ERQ | Up to six weeks prior to intervention, and again at 1 and 3 months post-intervention
  Emotion Regulation Questionnaire
DERS-18 | Up to six weeks prior to intervention, and again at 1 and 3 months post-intervention
  Difficulties in Emotion Regulation
PSQI | Up to six weeks prior to intervention, and again at 1 and 3 months post-intervention
  Pittsburgh Sleep Quality Index
IIP-32 | Up to six weeks prior to intervention, and again at 1 and 3 months post-intervention
  Inventory of Interpersonal Problems

CONTACTS AND LOCATIONS:
Locations (2):
- University of California, Berkeley, Berkeley, California, United States
- Bar-Ilan University, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be made available through the osf.io platform or similar platforms.